CLINICAL TRIAL: NCT00859027
Title: The Effect Of Risedronate On Bone Turnover And Bone Mass In Older Men
Brief Title: Effect Of Risedronate On Bone Mass In Older Men Receiving Neoadjuvant Therapy For Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Proctor and Gamble/Aventis (Unknown)
Responsible Party: Principal Investigator, Pamela Taxel, Principal Investigator, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-062; GCRC # 413; None given (Other Grant/Funding Number: Procotor and Gamble/Aventis); None given (Other: Procotor and Gamble/Aventis)
Record Dates: First submitted 2009-03-07; First posted 2009-03-10 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: Non-metastatic
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Risedronic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risedronate (Experimental): 35 mg by mouth every week as directed
  Interventions: Drug: risedronate
- risedronate placebo tablet (Placebo Comparator): Calcium and vitamin D
  Interventions: Drug: Placebo risedronate oral tablet

INTERVENTIONS:
Drug: risedronate — 35 mg/week by mouth
  Other Names: Actonel
  Arms: Risedronate
Drug: Placebo risedronate oral tablet — One tablet by mouth every week as directed
  Arms: risedronate placebo tablet

SUMMARY:
Men treated with neoadjuvant luteinizing hormone-releasing hormone (LHRH)-agonists such as leuprolide and goserelin for prostate cancer will become hypogonadal due to hormonal suppression and demonstrate increased bone turnover and consequent bone loss at the hip and spine. This bone loss can be prevented by treatment with 35 mg/week of risedronate.

DETAILED DESCRIPTION:
A 6-month randomized, double-blind, placebo-controlled trial was conducted, including 40 men aged ≥ 55 years receiving LHRH-agonist treatment for 6 months for locally advanced prostate cancer. Bone mineral density (BMD) of the lumbar spine, femoral neck, and total hip was measured every 6 months. In addition, bone turnover markers including N-telopeptide, serum C-telopeptide and procollagen peptide, and 25-OH vitamin D and intact parathyroid hormone were measured at baseline and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic prostate cancer
* Men to receive Gonadotropin-releasing Hormone-agonist therapy

Exclusion Criteria:

* Other cancers except skin cancer
* Evidence of metabolic bone disease
* Prior use of bisphosphonates

Ages: 55 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-01; Primary Completion 2008-03 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Taxel, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from medical clinics/ urology clinics.
Groups:
- Risedronate 35 mg p.o.Every Week Plus Calcium and Vit D Daily: Pts receiving LHRH-agonists for prostate cancer received active risedronate.
  They also received daily calcium + Vit D
- Calcium and Vitamin D Daily (Placebo Group): Pts received placebo risedronate + calcium and Vit D.
Period: Overall Study
Arm/Group | Risedronate 35 mg p.o.Every Week Plus Calcium and Vit D Daily | Calcium and Vitamin D Daily (Placebo Group)
Started | 25 | 25
Completed | 20 | 20
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risedronate Plus Calcium and Vit D | Calcium and Vitamin D | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (9) | 72 (7) | 71 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Mineral Density
Description: BMD was measured by dual-energy X-ray absorptiometry (Lunar DXA-IQ, Madison, WI, USA). The BMD of the femoral neck, total hip, and lumbar spine (L1-L4) was measured. Underlying data are no longer available; reported means have been estimated from the results publication.
Time Frame: baseline and 6 months
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Risedronate 35 mg p.o. Every Week Plus Calcium and Vit D Daily | Calcium and Vitamin D Daily (Placebo Group)
Number analyzed (Participants) | 20 | 20
Percent Change
  Femoral Neck | 0.1 (0.2) | -2 (0.5)
  Total Hip | 0.2 (0.3) | -2.2 (0.4)
  Lumbar Spine | 1.7 (0.8) | -1.3 (1)
Statistical Analysis 1: Comparison: Calcium and Vitamin D Daily (Placebo Group); Percent change in femoral neck BMD from baseline; Test type: Other; p = 0.004, One way ANOVA
Statistical Analysis 2: Comparison: Calcium and Vitamin D Daily (Placebo Group); Percent change in total hip BMD from baseline; Test type: Other; p = 0.001, One way ANOVA
Statistical Analysis 3: Comparison: Risedronate 35 mg p.o. Every Week Plus Calcium and Vit D Daily; Percent change in lumbar spine BMD from baseline; Test type: Other; p = 0.04, One way ANOVA
Statistical Analysis 4: Comparison: Risedronate 35 mg p.o. Every Week Plus Calcium and Vit D Daily vs Calcium and Vitamin D Daily (Placebo Group); Between group difference of percent change for the femoral neck BMD; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 5: Comparison: Risedronate 35 mg p.o. Every Week Plus Calcium and Vit D Daily vs Calcium and Vitamin D Daily (Placebo Group); Between group difference of percent change for total hip BMD; Test type: Other; p < 0.01, ANOVA

2. Secondary Outcome: Percent Change of Bone Turnover Markers
Description: Bone turnover markers including N-telopeptide (NTX), serum C-telopeptide (CTX) and procollagen peptide (P1NP), and 25-OH vitamin D and intact parathyroid hormone (PTH) were measured at baseline and at 6 months. Reported means have been estimated from the results publication as the underlying data are no longer available. Data for Vitamin D and PTH were not included in the publication.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Risedronate 35 mg p.o. Every Week Plus Calcium and Vit D Daily | Calcium and Vitamin D Daily (Placebo Group)
Number analyzed (Participants) | 20 | 20
Percent Change
  NTX | -15 (3) | 21 (2)
  CTX | -5 (4) | 55 (5)
  P1NP | -1 (2) | 41 (4)
  Vitamin D | NA (NA) — Underlying data not available | NA (NA) — Underlying data not available
  PTH | NA (NA) — Underlying data not available | NA (NA) — Underlying data not available
Statistical Analysis 1: Comparison: Risedronate 35 mg p.o. Every Week Plus Calcium and Vit D Daily vs Calcium and Vitamin D Daily (Placebo Group); Between group difference of percent change for NTX; Test type: Other; p = 0.015, ANOVA
Statistical Analysis 2: Comparison: Risedronate 35 mg p.o. Every Week Plus Calcium and Vit D Daily vs Calcium and Vitamin D Daily (Placebo Group); Between group difference of percent change for CTX; Test type: Other; p = 0.01, ANOVA

ADVERSE EVENTS:
Groups:
- Risedronate: Particiapnts given 35 mg by mouth every week
Arm/Group | Calcium and Vitamin D | Risedronate
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Small number but otherwise no limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes